CLINICAL TRIAL: NCT00245479
Title: An Open Label, Multi-national Study of Oral Desmopressin in Previously Untreated Children Aged 5 to 15 Years With Primary Nocturnal Enuresis
Brief Title: A Study of Oral Desmopressin in Previously Untreated Children Aged 5 to 15 Years With Primary Nocturnal Enuresis
Acronym: DRIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE992026 CS002
Record Dates: First submitted 2005-09-13; First posted 2005-10-28 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Nocturnal Enuresis
Keywords: Primary nocturnal enuresis
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Primary nocturnal enuresis

INTERVENTIONS:
Drug: Primary nocturnal enuresis — Desmopressin

SUMMARY:
To evaluate the overall response to desmopressin treatment among previously untreated enuretic children aged 5-15 years after 3 and 6 months of treatment.

To investigate the influence of possible predictive factors on response after 3 and 6 months of treatment.

To evaluate the proportion of patients achieving dryness. To evaluate the long-term safety profile of oral desmopressin in children with primary nocturnal enuresis.

DETAILED DESCRIPTION:
To evaluate the overall response to desmopressin treatment among previously untreated enuretic children aged 5-15 years after 3 and 6 months of treatment.

To investigate the influence of possible predictive factors on response after 3 and 6 months of treatment.

To evaluate the proportion of patients achieving dryness. To evaluate the long-term safety profile of oral desmopressin in children with primary nocturnal enuresis.

ELIGIBILITY:
Inclusion criteria:

* Children suffering from primary nocturnal enuresis with no organic pathology.
* Children of either sex, not below 5 and not above 15 years of age (not below 6 years in The Netherlands and France).
* Children with a minimum of 6 wet nights in 2 weeks.

Exclusion criteria:

* Children who have previously been treated with desmopressin or other medications for nocturnal enuresis or enuresis alarms.
* Children receiving substances that are known or suspected to potentiate antidiuretic hormone, e.g. SSRI, tricyclic antidepressant drugs, chlorpromazine and carbamazepine.
* Diagnosed renal diabetes insipidus or central diabetes insipidus with an AVP (arginine vasopressin) deficiency.
* Proven urinary tract infection within the past month or a documented positive urine culture at the start of the study

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 802 (Actual)
Dates: Start 2002-04; Primary Completion 2005-09 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall response to desmopressin treatment among previously untreated enuretic children aged 5-15 years after 3 and 6 months of treatment

SECONDARY OUTCOMES:
To investigate the influence of possible predictive factors on response after 3 and 6 months of treatment.
To evaluate the proportion of patients achieving dryness.
To evaluate the long-term safety profile of oral desmopressin in children with primary nocturnal enuresis.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Foundation Hospital Saint Joseph, 185, rue Raymond Losserand, Paris, France

REFERENCES:
- [Derived] Van Herzeele C, Evans J, Eggert P, Lottmann H, Norgaard JP, Vande Walle J. Predictive parameters of response to desmopressin in primary nocturnal enuresis. J Pediatr Urol. 2015 Aug;11(4):200.e1-8. doi: 10.1016/j.jpurol.2015.03.007. Epub 2015 May 21. PMID 26059526
- [Derived] Van Herzeele C, De Bruyne P, Evans J, Eggert P, Lottmann H, Norgaard JP, Vande Walle J. Safety profile of desmopressin tablet for enuresis in a prospective study. Adv Ther. 2014 Dec;31(12):1306-16. doi: 10.1007/s12325-014-0173-1. Epub 2014 Dec 12. PMID 25504157
- [Derived] Lottmann H, Baydala L, Eggert P, Klein BM, Evans J, Norgaard JP. Long-term desmopressin response in primary nocturnal enuresis: open-label, multinational study. Int J Clin Pract. 2009 Jan;63(1):35-45. doi: 10.1111/j.1742-1241.2008.01956.x. PMID 19125991